CLINICAL TRIAL: NCT01931332
Title: Randomised, Observer Blinded, Controlled Trial of Intrathecal Diamorphine Versus Femoral Nerve Block for Post-operative Analgesia Following Primary Total Knee Arthroplasty
Brief Title: Intrathecal Diamorphine Versus Femoral Nerve Block in Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Matthew Grayling, Consultant Anaesthetist, Royal Devon and Exeter NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10/H0202/1
Record Dates: First submitted 2013-08-20; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; Analgesia
MeSH Terms: conditions — Osteoarthritis; Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Nerve Block with levobupivicaine (Active Comparator): A single injection femoral nerve block (FNB) was performed in the supine position with a 50mm insulated needle (NanoLine, Pajunk, Geisingen, Germany) and peripheral nerve stimulator set at 1Hertz (Hz) with pulse width 0.1ms. Once a quadriceps muscle twitch was identified at a stimulated current between 0.2 and 0.5milliamperes (mA), 20mls of 0.375% levobupivacaine (75mg) was injected in fractionated amounts after negative aspiration
  Interventions: Procedure: Femoral Nerve Block with levobupivicaine
- Intrathecal injection of diamorphine (Active Comparator): 500mcg of intrathecal diamorphine (ID) (dissolved in 0.5mls normal saline)
  Interventions: Procedure: Intrathecal injection of diamorphine

INTERVENTIONS:
Procedure: Femoral Nerve Block with levobupivicaine — A single injection femoral nerve block (FNB) performed in the supine position with a 50mm insulated needle (NanoLine, Pajunk, Geisingen, Germany) and peripheral nerve stimulator set at 1Hz with pulse width 0.1ms. Once a quadriceps muscle twitch is identified at a stimulated current between 0.2 and 0.5mA, 20mls of 0.375% levobupivacaine (75mg) is injected in fractionated amounts after negative aspiration
  Arms: Femoral Nerve Block with levobupivicaine
Procedure: Intrathecal injection of diamorphine — 500mcg of intrathecal diamorphine (ID) (dissolved in 0.5mls normal saline)
  Arms: Intrathecal injection of diamorphine

SUMMARY:
Primary total knee arthroplasty (TKA) is commonly associated with moderate to severe early post-operative pain. The primary aim of this study was to investigate the impact of either a single-shot femoral nerve block (FNB) or intrathecal diamorphine (ID) on post-operative pain after TKA

The Null Hypothesis is that there is no difference in the post operative pain relief provided for TKA by a single-shot femoral nerve block (FNB) as compared to intrathecal diamorphine (ID).

DETAILED DESCRIPTION:
In 2008, the Prospect Working Group, a multidisciplinary expert panel, published their consensus guidelines on the relative merits of different anaesthetic and analgesic techniques for TKA based on a review of the available published literature up to 2005. These guidelines supported the use of general anaesthesia combined with a femoral nerve block for surgery and postoperative analgesia, or alternatively spinal anaesthesia with local anaesthetic combined with spinal morphine. The preference for femoral nerve block in favour of intrathecal opiates was as a consequence of the greater potential for side effects with the latter technique. The authors conceded that there were a lack of well-conducted studies on this subject, graded their recommendations as level D (expert opinion), and concluded further research was needed. Consequently there has been debate around the conclusions drawn and clinicians have not universally accepted the recommendations.

Most researchers to date have focused on short-term outcomes such as static pain scores and/or opiate consumption. It is also important however to investigate dynamic pain scores, patient reported outcomes, the attainment of rehabilitation goals, length of stay and longer term functional outcomes. In addition, the use of the total pain relief score (TOTPAR) as described by Cooper and Beaver, assesses the cumulative response to treatment. This is a well validated area under the time-analgesic effect curve (AUC) derivation for pain relief which is commonly used by meta-analyses of analgesic interventions. The aim of this study is to investigate all these endpoints in patients receiving a single-shot femoral nerve block (FNB) for TKA as compared to intrathecal diamorphine (ID), a more commonly used spinal opiate in United Kingdom anaesthetic practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for primary unilateral Total Knee Arthroplasty

Exclusion Criteria:

* Uni-compartmental surgery, bilateral surgery, contra-indication to spinal anaesthesia or peripheral nerve block (anticoagulation, hydrocephalus, raised intracranial pressure), allergy to local anaesthetics or diamorphine, malignant hyperthermia or other concerns over general anaesthesia, chronic opiate use and chronic pain medication use (e.g. gabapentin, pregabalin, amitriptyline).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Median pain score (NRS: see below) at rest | Over 72 hours post operatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain) assessed at times 3, 6, 12, 24, 48 and 72 hrs postoperatively.

SECONDARY OUTCOMES:
Pain on movement | At 3 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain on movement | At 6 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain on movement | At 12 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain on movement | At 24 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain on movement | At 48 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain on movement | At 72 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain at rest | At 3 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain at rest | At 6 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain at rest | At 12 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain at rest | At 24 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain at rest | At 48 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Pain at rest | At 72 hrs postoperatively
  Numerical rating scale (NRS) score (where 0 = no pain and 10 = worst possible pain)
Morphine consumption | Over 72 hrs postoperatively
  Cumulative consumption in milligrams

OTHER OUTCOMES:
Quality of recovery score 40 | Day 2 post operatively
  Quality of recovery score is a 40 point patient reported outcome measure devised by Paul Myles and reported in the British Journal of Anaesthesia 84 (1): 11-15 (2000). This psychometric tool assess emotional state, physical comfort, psychological support, physical independence and pain grading each out of 5 (0= lowest score and 5 = highest score). We ranked total score as extremely poor (0-40), poor (41-80), satisfactory (81-120), good (121-160) or excellent (161-200).
Total Pain Relief Score (TOTPAR) | Day 1,2 and 3 post-operatively
  Percentage of the maximum total pain relief was calculated by dividing the total pain relief (TOTPAR) over the three days by the maximum potential pain relief and expressed as a percentage (%maxTOTPAR)
Functional health outcome measure | At 6 weeks post-operatively
  The Oxford Knee Score (OKS) is a 12-item patient-reported questionnaire specifically designed and developed to assess function and pain after total knee arthroplasty. It is short, reproducible, valid and sensitive to clinically important changes.
  The OKS was designed to be completed by the patient thus minimising potential bias unwittingly introduced by surgeons when assessing the results themselves.
  The PRO was designed and developed by researchers within Public Health and Primary Health Care at the University of Oxford in association with surgical colleagues at the Nuffield Orthopaedic Centre.
  The OKS at 6 weeks was compared to the preoperative OKS to describe the change in functional outcome.
Physical health outcome | A 6 weeks post-operatively
  EuroQol 5 Dimensions Score/Visual Analogue Score (EQ-5D™/VAS). This is a standardised instrument for use as a measure of health outcome. It uses a patient self reporting 5 point (3 level) questionnaire and visual analogue scale to measure health. Health improvement at 6 weeks was assessed by comparing with pre-operative scores.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Grayling, MBBS, Principal Investigator — Royal Devon and Exeter Hospital
Locations (1):
- Royal Devon and Exeter Hospital, Exeter, Devon, United Kingdom